CLINICAL TRIAL: NCT04063774
Title: Multicenter Clinical Trial of the Validity and Impact of Diagnostic Tests and Clinical Algorithms for Dengue in Febrile Subjects in Endemic Areas in Colombia 2016
Brief Title: Clinical Trial of Diagnostic Tests and Clinical Algorithms for Dengue in Febrile Subjects in Endemic Areas in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lyda Osorio (Other)
Collaborators: COMFANDI CAJA DE COMPENSACION DEL VALLE DEL CAUCA (Unknown); SISTEMA GENERAL DE REGALIAS CASANARE, SANTANDER VALLE DEL CAUCA (Unknown); RED AEDES (Unknown)
Responsible Party: Sponsor-Investigator, Lyda Osorio, Professor, Universidad del Valle, Colombia
Organization: Universidad del Valle, Colombia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 144-016
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Dengue
Keywords: diagnostics; sensitivity; specificity; clinical algorithm
MeSH Terms: conditions — Dengue; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Algorithms were developed and validated in silico, those with the highest sensitivity were tested in consecutive eligible subjects and their performance compared to dengue reference tests (gold standard combination of tests). Algorithms were modified according to intermediate analysis of performance planned in advance
Masking Description: Samples were coded and laboratory personnel were unaware of algorithm results, the participant did not know what algorithm prototype was tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dengue diagnostic algorithm (Experimental): single arm of consecutive enrolled subjects with fever in whom the dengue diagnostic algorithms were applied by study physician and blood sample taken for hemogram and dengue reference tests (gold standard)
  Interventions: Diagnostic Test: Dengue calculator

INTERVENTIONS:
Diagnostic Test: Dengue calculator — Clinical diagnostic algorithms of dengue generated by discrete and continuos Bayes formulas installed in a mobile device

SUMMARY:
The present study aimed to develop a sensitive dengue diagnostic clinical algorithm using the resources that are available at the health care institutions, clinical expertise, and identification of signs and symptoms and variables of the hemogram associated with dengue. The performance of the potential algorithms were assessed under routine care. A single group cuasiexperimental study with a Bayesian adaptive design was conducted. Prior and cumulative information was used during intermediate analysis of clinical algorithms performance and according to these results algorithms were modified and then implemented in the subsequent study subjects. Men and women of all ages, seeking care due to fever of less than 15 days were recruited in 3 endemic areas in Colombia. The algorithms were applied by study physicians and blood samples taken for hemogram and dengue reference tests. It was planned that algorithms with high sensitivity (95%) and specificity (80%) were implemented in real life to assess their impact on patients outcomes alone and in combination with dengue rapid diagnostic tests but this was not feasible as not algorithms achieved the targetted performance. The experience of physicians using the algorithm in a mobile device was going to be explored with qualitative methods but this was explored with study physicians.

ELIGIBILITY:
Inclusion Criteria:

* Fever of less than 15 days

Exclusion Criteria:

* Origin of fever identified

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of dengue calculator | 0 days
  Number of correctly identified dengue cases by intervention out of all laboratory confirmed dengue cases
Specificity of dengue calculator | 0 days
  Number of correctly identified non-dengue cases by intervention out of all laboratory confirmed non-dengue cases

SECONDARY OUTCOMES:
Sensitivity in dengue and probable dengue cases | 0 days
  Number of correctly identified dengue cases by intervention out of all laboratory confirmed plus probable dengue cases

CONTACTS AND LOCATIONS:
Overall Officials: Lyda Osorio, MD PhD, Principal Investigator — Universidad del Valle; Diana Ma Caicedo, MD MSc, Principal Investigator — Universidad del Valle
Locations (3):
- Colombia (3):
  - Hospital Regional de la Orinoquía, Yopal, Casanare Department
  - Clinica y Hospital Local de Piedecuesta, Piedecuesta, Santander Department
  - COMFANDI Torres y Alameda, Cali, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: Yes
Patient unidentifiable data and detailed algorithms available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request for 10 years